CLINICAL TRIAL: NCT00678392
Title: AXITINIB (AG-013736) AS SECOND LINE THERAPY FOR METASTATIC RENAL CELL CANCER: AXIS TRIAL
Brief Title: Axitinib (AG 013736) As Second Line Therapy For Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4061032; AXIS TRIAL; 2008-001451-21 (EudraCT Number); AXIS (Other: Alias Study Number)
Record Dates: First submitted 2008-05-12; First posted 2008-05-15 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Kidney Neoplasms
Keywords: Axitinib in Second Line Treatment of Patients With Metastatic Renal Cell Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Axitinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Axitinib (Experimental)
  Interventions: Drug: Axitinib (AG-013736)
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Axitinib (AG-013736) — axitinib will be given at a starting dose of 5 mg twice daily [BID] with continuous dosing
  Arms: Axitinib
Drug: Sorafenib — sorafenib will be given at a dose of 400 mg twice daily [BID] with continuous dosing
  Arms: Sorafenib

SUMMARY:
The study is designed to demonstrate that axitinib (AG-013736) is superior to sorafenib in delaying tumor progression in patients with metastatic renal cell cancer after failure of one first line regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell cancer with a component of clear cell subtype, with metastasis
* Evidence of measurable disease
* Must have failed one prior systemic first-line regimen for metastatic renal cell cancer

Exclusion Criteria:

* Prior treatment for metastatic renal cell cancer with more that one systemic first line therapy
* Major surgery less than 4 weeks or radiation less than 2 weeks of starting study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2008-09-03 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2016-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (281):
- United States (148):
  - East Valley Hematology and Oncology Medical Group, Burbank, California
  - Maurice Berkowtiz, MD, Burbank, California
  - Agajanian Institute of Oncology and Hematology, Downey, California
  - Los Angeles Hematology/Oncology Medical Group, Glendale, California
  - Los Angeles Hematology/Oncology Medical Group, Los Angeles, California
  - LAC-USC Medical Center, Los Angeles, California
  - USC Norris Cancer Hospital and Clinics, Los Angeles, California
  - Kenmar Research Institute, Los Angeles, California
  - Metropolitan Hematology/Oncology Medical Group, Los Angeles, California
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Agajanian Institute of Oncology and Hematology, Montebello, California
  - Brian LeBerthon, MD, A Medical Corporation, West Covina, California
  - Agajanian Institute of Oncology and Hematology, Whittier, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Denver: Division of Medical Oncology, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Georgetown University Hospital, Lombardi Cancer Center, Washington D.C., District of Columbia
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - University of Miami Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - Florida Cancer Specialists, Englewood, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - Florida Cancer Specialists, Naples, Florida
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Peachtree Hematology-Oncology Consultants, P.C., Atlanta, Georgia
  - Chattanooga Oncology and Hematology Associates, PC, Ringgold, Georgia
  - Mountain States Tumor Institute, Boise, Idaho
  - Mountain States Tumor Institute, Fruitland, Idaho
  - Mountain States Tumor Institute, Meridian, Idaho
  - Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute, Twin Falls, Idaho
  - Loyola University Chicago Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Cental Indiana Cancer Centers, Carmel, Indiana
  - Central Indiana Cancer Centers, Fishers, Indiana
  - Cental Indiana Cancer Centers, Greenfield, Indiana
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - St. John's Mercy, David C. Pratt Cancer Center, St Louis, Missouri
  - St. John's Mercy Medical Center, Washington, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Center at Hackensack University Medical Center - The Hillcrest Building, Hackensack, New Jersey
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center - Sidney Kimmel Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Department of Medicine MSG @ SUNY HSC @ Syrcacuse, Inc., Oneida, New York
  - Department of Medicine MSG @ SUNY HSC @ Syracuse, Inc., Oswego, New York
  - Suny Upstate Medical University, Syracuse, New York
  - Department of Medicine MSG @ SUNY HSC @ Syracuse, Inc, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Raleigh Hematology Oncology Associates, DBA, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Investigational Chemotherapy Services, Durham, North Carolina
  - Albermarie Hospitals, Elizabeth City, North Carolina
  - Virginia Oncology Associates, Elizabeth City, North Carolina
  - Raleigh Hematology Oncology Associates, P.C., Raleigh, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Arthur G. James Cancer Hospital and Richard J. Solove Research Institute, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - James Care in Kenny, Columbus, Ohio
  - Monarch, Mayfield Heights, Ohio
  - Lake University - Ireland Cancer Center (LUICC), Mentor, Ohio
  - UHHS - Chagrin Highlands, Orange, Ohio
  - UHHS - Westlake, Westlake, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas, Easley, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Hematology and Oncology Associates of SC, LLC - Eastside Medical Center, Greenville, South Carolina
  - Cancer Centers of the Carolinas, Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas, Spartanburg, South Carolina
  - Chattanooga Oncology and Hematology Associates, PC, Chattanooga, Tennessee
  - Chattanooga Oncology Hematology Associates P.C., Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center-Cool Springs, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Chattanooga Oncology & Hematology Associates, Hixson, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Central Midtown, Austin, Texas
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncolgoy - Austin North, Austin, Texas
  - Texas Oncology - Austin Northwest, Austin, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Oncology - Cedar Park, Cedar Park, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Investigation Products Center (IPC), Fort Worth, Texas
  - Investigational Products Center (IPC), Fort Worth, Texas
  - US Oncology Research and Clinical Pharmacy, Fort Worth, Texas
  - Genitourinary Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock, Round Rock, Texas
  - Texas Oncology, P.A., Tyler, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology - Clear Lake, Webster, Texas
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Virginia Cancer Specialists, PC, Woodbridge, Virginia
  - Virginia Mason Medical Center, Section of Hematology/Oncology, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (6):
  - The Canberra Hospital, Medical Oncology, Garran, Australian Capital Territory
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Ballarat Oncology & Haematology Services, Ballarat, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Hospital, Austin Health, Heidelberg, Victoria
  - Heidelberg Repatriation Hospital, Austin Health, Heidelberg West, Victoria
- Austria (2):
  - Med. Abt. KH Barmherzige Brueder Wien, Krankenhaus der Barmherzigen Brueder Wien, Vienna
  - Universitaets-Klinik fuer Innere Medizin I, Vienna
- Brazil (4):
  - Clinica Oncologistas Associados, Rio de Janeiro, Rio de Janeiro
  - Irmandade da Santa Casa de Misericordia de Porto Alegre (ISCMPA) - Hospital Santa Rita, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Fundacao Antonio Prudente, São Paulo, São Paulo
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - RSM Durham Regional Cancer Centre Lakeridge Health Oshawa, Oshawa, Ontario
- China (7):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Chaoyang District
  - The Department of Medical Oncology, PLA Cancer Center, Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Beijing Cancer Hospital, Beijing, P.R.
  - Xijing Hospital, The Fourth Military Medical University, Xi'an, Shaanxi
  - Sun Yet-Sen University Cancer Center, Guangzhou
  - Urology Department, Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tianjin Oncology Hospital,biology treatment department, Tianjin
- France (10):
  - Centre Leon Berard, Lyon, Cedex 08
  - Hopital Saint-André, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - Institut Paoli-Calmettes, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Rene Gauducheau - Service Oncologie Medicale, Saint-Herblain
  - CHRU de Tours - Hopital Bretonneau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy / Service d'Immunotherapie, Villejuif
- Germany (7):
  - RWTH Aachen, Urologische Klinik, Aachen
  - Charite - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Innere Klinik und Poliklinik fuer Tumorforschung, Universitaetsklinikum Essen, Essen
  - Klinikum Region Hannover Krankenhaus Siloah, Hanover
  - Klinikum der Johannes-Gutenberg-Universitaet, III. Medizinische Klinik und Poliklinik, Mainz
  - Ludwig-Maximilians-Universitaet Muenchen, Klinikum Grosshadern Urologische Klinik und Poliklinik, München
  - Klinikum Oldenburg gGmbH, Klinik fuer Innere Medizin II Onkologie / Haematologie, Oldenburg
- Greece (2):
  - Alexandra University Hospital / Oncology Dept., Athens, Attica
  - "Theagenio"Cancer Hospital / 3rd. Dept. of Clinical Oncology, Thessaloniki, Macedonia
- India (5):
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Dept. of Medical Oncology, Tata Memorial Hospital, Mumbai, Maharashtra
  - Christian Medical College & Hospital, Ludhiana, Punjab
  - Bhagwan Mahaveer Cancer Hospital and Research Center, Jaipur, Rajasthan
- Oncology Department, Dublin, Ireland
- Italy (14):
  - UOC Oncologia Medica, Ospedale San Donato, Arezzo
  - Centro di Riferimento Oncologico, Istituto Nazionale Tumori, IRCCS, Aviano (PN)
  - Dipartimento dei laboratori diagnositici e per le terapie cellulari, Aviano (PN)
  - Azienda Ospedaliera Spedali Civili di Brescia, Unita' Operativa Oncologia Medica, Brescia
  - Struttura Complessa di Oncologia, Cremona
  - UOC Oncologia Medica B, IRCCS AO Universitaria San Martino, Genova
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, SC Oncologia Medica 2, Milan
  - Divisione di Oncologia, AORN Antonio Cardarelli, Napoli
  - Istituto per lo Studio e la Cura dei Tumori Fondazione Pascale, Napoli
  - Unita' Operativa Oncologia Medica 2, Regione del Veneto, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Struttura Complessa di Oncologia Medica A, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Oncologia Medica, Padiglione Flajani, I piano, Roma
  - UO di Oncologia ed Ematologia, Istituto Clinico Humanitas, Rozzano (MI)
- Japan (18):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo Medical University School of Medicine, Sapporo, Hokkaido
  - University of Tsukuba, Graduate School of Comprehensive Human Sciences, Department of Urology, Tsukuba, Ibaraki
  - Kinki University Hospital, Sayama, Osaka
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Tokyo Women's Medical University Medical Center East, Department of Urology, Arakawa-ku, Tokyo
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
  - Akita University Hospital, Akita
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Kumamoto University Hospital, Kumamoto
  - Tokushima University, Tokushima
  - Yamagata University Hospital, Yamagata
- Poland (7):
  - Centrum Medyczne HCP, Poznan, Wielkopolska
  - Wielkopolskie Centrum Onkologii im.Marii Sklodowskiej-Curie, Poznan, Wielkopolska
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Klinika Onkologii, Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego, Poznan
  - Pracownia Tomografii Komputerowej, Poznan
  - Klinika Onkologii, Wojskowy Instytut Medyczny, Warsaw
  - Klinika Urologii i Onkologii Urologicznej, Wroclaw
- Russia (7):
  - Medical Radiology Research Center of the Minzdravsotsrazvitiya of Russia, Obninsk, Kaluga Oblast
  - Cancer Research Center named after N.N. Blokhin, Biotherapy Department, Moscow
  - Cancer Research Center named after N.N.Blokhin, Chemotherapy Department, Moscow
  - Russian Research Center of Roentgenology and Radiology, Moscow
  - The Main Clinical Hospital of the Ministry of Internal Affairs of Russian Federation, Moscow
  - Moscow Research Institute of Oncology P.A. Herzen, Moscow
  - City Clinical Oncology Dispensary, Saint Petersburg
- National Cancer Centre Singapore, Singapore, Singapore
- Slovakia (3):
  - Onkologicky Ustav sv. Alzbety, Bratislava
  - Narodny Onkologicky ustav, Bratislava
  - Nemocnica s poliklinikou Zilina, Žilina
- South Korea (6):
  - National Cancer Center, Urologic Oncology Clinic, Center for Specific Organs Cancer, Goyang-si, Gyeonggi-do
  - Dong-A University Medical Center, Department of Medicine, Division of Hemato-Oncology, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Catholic University of Korea, Seoul St. Mary's Hospital, Department of Oncology, Seoul
- Spain (9):
  - Institut Catala D'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Vall D¿Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Universitetssjukhuset, Onkologiska kliniken, Linköping
  - Norrlands Universitetssjukhus, Onkologkliniken, Umeå
  - Onkologkliniken, Vaxjo
- Taiwan (4):
  - Chang Gung Medical Foundation-Kaohsiung Branch, Kaohsiung Hsien
  - Taichung Veterans General Hospital, Department of Surgery, Taichung
  - Department of Oncology, National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (11):
  - Royal Marsden Hospital, London, England
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Clatterbridge Centre for Oncology NHS Foundation Trust, Bebington, Wirral
  - University of Birmingham, CRUK Institute for Cancer Studies, Birmingham
  - Royal Bournemouth & Poole Hospitals, Bournemouth
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Department of Medical Oncology, St. Bartholomew's Hospital, London
  - University Department of Medical Oncology/Oxford Cancer Centre, Oxford
  - Royal Marsden Hospital NHS Foundation Trust, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Rini BI, Atkins MB, Choueiri TK, Teresi RE, Rosbrook B, Thakur M, Hutson TE. Plain language summary looking at how long side effects last after treatment with axitinib is stopped in people with advanced renal cell carcinoma. Future Oncol. 2023 Dec;19(40):2623-2629. doi: 10.2217/fon-2023-0233. Epub 2023 Aug 1. PMID 37526095
- [Derived] Murphy DA, Rini BI, Escudier B, Motzer RJ, Wang P, Li S, Williams JA, Tarazi JC, Martini JF. Angiogenic and immunomodulatory biomarkers in axitinib-treated patients with advanced renal cell carcinoma. Future Oncol. 2020 Jun;16(17):1199-1210. doi: 10.2217/fon-2020-0212. Epub 2020 May 4. PMID 32363929
- [Derived] Bracarda S, Bamias A, Casper J, Negrier S, Sella A, Staehler M, Tarazi J, Felici A, Rosbrook B, Jardinaud-Lopez M, Escudier B. Is Axitinib Still a Valid Option for mRCC in the Second-Line Setting? Prognostic Factor Analyses From the AXIS Trial. Clin Genitourin Cancer. 2019 Jun;17(3):e689-e703. doi: 10.1016/j.clgc.2019.03.017. Epub 2019 Apr 1. PMID 31072748
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- [Derived] Escudier B, Michaelson MD, Motzer RJ, Hutson TE, Clark JI, Lim HY, Porfiri E, Zalewski P, Kannourakis G, Staehler M, Tarazi J, Rosbrook B, Cisar L, Hariharan S, Kim S, Rini BI. Axitinib versus sorafenib in advanced renal cell carcinoma: subanalyses by prior therapy from a randomised phase III trial. Br J Cancer. 2014 Jun 10;110(12):2821-8. doi: 10.1038/bjc.2014.244. Epub 2014 May 13. PMID 24823696
- [Derived] Ueda T, Uemura H, Tomita Y, Tsukamoto T, Kanayama H, Shinohara N, Tarazi J, Chen C, Kim S, Ozono S, Naito S, Akaza H. Efficacy and safety of axitinib versus sorafenib in metastatic renal cell carcinoma: subgroup analysis of Japanese patients from the global randomized Phase 3 AXIS trial. Jpn J Clin Oncol. 2013 Jun;43(6):616-28. doi: 10.1093/jjco/hyt054. Epub 2013 Apr 28. PMID 23630366
- [Derived] Motzer RJ, Escudier B, Tomczak P, Hutson TE, Michaelson MD, Negrier S, Oudard S, Gore ME, Tarazi J, Hariharan S, Chen C, Rosbrook B, Kim S, Rini BI. Axitinib versus sorafenib as second-line treatment for advanced renal cell carcinoma: overall survival analysis and updated results from a randomised phase 3 trial. Lancet Oncol. 2013 May;14(6):552-62. doi: 10.1016/S1470-2045(13)70093-7. Epub 2013 Apr 16. PMID 23598172
- [Derived] Cella D, Escudier B, Rini B, Chen C, Bhattacharyya H, Tarazi J, Rosbrook B, Kim S, Motzer R. Patient-reported outcomes for axitinib vs sorafenib in metastatic renal cell carcinoma: phase III (AXIS) trial. Br J Cancer. 2013 Apr 30;108(8):1571-8. doi: 10.1038/bjc.2013.145. Epub 2013 Apr 11. PMID 23579211
- [Derived] Rini BI, Escudier B, Tomczak P, Kaprin A, Szczylik C, Hutson TE, Michaelson MD, Gorbunova VA, Gore ME, Rusakov IG, Negrier S, Ou YC, Castellano D, Lim HY, Uemura H, Tarazi J, Cella D, Chen C, Rosbrook B, Kim S, Motzer RJ. Comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS): a randomised phase 3 trial. Lancet. 2011 Dec 3;378(9807):1931-9. doi: 10.1016/S0140-6736(11)61613-9. Epub 2011 Nov 4. PMID 22056247

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib 5 mg: Axitinib (AG-013736) 5 milligram (mg) tablet administered orally twice daily in cycles of 4 weeks.
- Sorafenib 400 mg: Sorafenib 400 mg tablet administered orally twice daily in cycles of 4 weeks.
Period: Overall Study
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Started | 361 | 362
Treated | 359 | 355
Completed | 0 | 0
Not Completed | 361 | 362
Not completed — Adverse Event | 0 | 6
Not completed — Death | 280 | 269
Not completed — Lost to Follow-up | 15 | 13
Not completed — Objective Progression or Relapse | 3 | 8
Not completed — Sponsor's Decision | 1 | 2
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Randomized But Not Treated | 2 | 7
Not completed — Other | 56 | 53

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or receive a different drug from that to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg | Total
Number analyzed (Participants) | 361 | 362 | 723
Age, Customized [Number; unit: Participants]
  Less than (<) 65 years | 238 | 238 | 476
  Greater than or equal to (>=) 65 years | 123 | 124 | 247
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 104 | 200
  Male | 265 | 258 | 523

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time in months from start of study treatment to the first documentation of objective tumor progression of disease (PD) or to death due to any cause, whichever occurs first. PD was assessed by response evaluation criteria in solid tumors (RECIST) version 1.0. PD: >=20 percent (%) increase in the sum of the longest dimensions (LD) of the target lesions taking as a reference the smallest sum of the LD recorded since the start of treatment or unequivocal progression in non-target lesions or the appearance of 1 or more new lesions. Occurrence of a pleural effusion or ascites was also considered PD if demonstrated by cytological investigation and it was not previously documented. New bone lesions not previously documented were considered PD if confirmed by computed tomography/magnetic resonance imaging or X-ray.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: FAS included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Months | 6.7 [6.3 to 8.6] | 4.7 [4.6 to 5.6]
Statistical Analysis 1: Comparison: Axitinib 5 mg vs Sorafenib 400 mg; Test type: Superiority or Other; p < 0.0001, Log Rank — P-value was obtained from 1-sided log rank test, stratified by eastern cooperative oncology group (ECOG) and prior treatment. One-sided log-rank test at 0.025 level of significance was used to compare PFS between the 2 treatment arms; Hazard Ratio (HR) = 0.665, 95% CI 2-sided [0.544 to 0.812]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from start of study treatment to date of death due to any cause. OS was calculated as (months) = (date of death minus the date of first dose of study medication plus 1) divided by 30.4. For participants who were alive, overall survival was censored on last date the participants were known to be alive.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Months | 20.1 [16.7 to 23.4] | 19.2 [17.5 to 22.3]
Statistical Analysis 1: Comparison: Axitinib 5 mg vs Sorafenib 400 mg; Test type: Superiority or Other; p = 0.3744, Log Rank; P-value was obtained from a 1-sided log-rank test of treatment stratified by ECOG performance status and prior treatment; Hazard Ratio (HR) = 0.969, 95% CI 2-sided [0.800 to 1.174]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR = percentage of participants with confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.0 recorded from first dose of study treatment until PD or death due to any cause. CR: disappearance of all target, non target lesions and no appearance of new lesions, documented on 2 occasions separated by at least 4 weeks. PR: at least 30 % decrease in sum of LD of target lesions taking as reference baseline sum of LD, without progression of non target lesions, no appearance of new lesions. PD: >=20% increase in sum of LD of the target lesions taking as a reference smallest sum of LD recorded since the start of treatment or unequivocal progression in non-target lesions or appearance of 1 or more new lesions. Occurrence of pleural effusion or ascites if demonstrated by cytological investigation, not previously documented. New bone lesions not previously documented if confirmed by computed tomography/magnetic resonance imaging or X-ray.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Percentage of participants | 19.4 [15.4 to 23.9] | 9.4 [6.6 to 12.9]
Statistical Analysis 1: Comparison: Axitinib 5 mg vs Sorafenib 400 mg; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; P-value was obtained from a 1-sided Cochran-Mantel-Haenszel test of treatment stratified by ECOG performance status and prior treatment; Risk Ratio (RR) = 2.056, 95% CI 2-sided [1.408 to 3.003]

4. Secondary Outcome: Duration of Response (DR)
Description: DR: time from first documentation of objective tumor response (CR or PR), that was subsequently confirmed, to the first documentation of PD or to death due to any cause, whichever occurred first as per RECIST version 1.0, a) CR: disappearance of all target, non target lesions and no appearance of new lesions, documented on 2 occasions separated by at least 4 weeks, b) PR: at least 30 % decrease in sum of LD of target lesions taking as reference baseline sum of LD, without progression of non target lesions, no appearance of new lesions, c) PD: >=20% increase in sum of LD of the target lesions taking as a reference smallest sum of LD recorded since the start of treatment or unequivocal progression in non-target lesions or appearance of 1 or more new lesions. Occurrence of pleural effusion or ascites if demonstrated by cytological investigation, not previously documented. New bone lesions not previously documented if confirmed by computed tomography/magnetic resonance imaging or X-ray.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Months | 11.0 [7.4 to NA] — The upper limit of 95 percent confidence interval was not reached at the time of data cut-off. | 10.6 [8.8 to 11.5]

5. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life- threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: Safety population included all participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 359 | 355
Percentage of participants
  AEs | 96.1 | 98.0
  SAEs | 40.7 | 35.8

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of the AEs was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Grade 1= mild; Grade 2= moderate; Grade 3= severe; Grade 4= life-threatening or disabling; Grade 5= death related to AE.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 359 | 355
Percentage of participants
  Grade 1 | 3.9 | 3.1
  Grade 2 | 20.1 | 21.7
  Grade 3 | 47.6 | 52.4
  Grade 4 | 10.6 | 11.5
  Grade 5 | 13.9 | 9.3

7. Secondary Outcome: Percentage of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life -threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious and non -serious AEs.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 359 | 355
Percentage of participants
  AEs | 92.2 | 95.2
  SAEs | 15.3 | 13.8

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Hematology
Description: Hematology laboratory test included hemoglobin, platelet count, white blood cells count, neutrophils and lymphocytes. Abnormalities were assessed by CTCAE Grade Version 2 for severity: Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: Safety population included all participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received. Here, "n" signifies number of participants available for specified categories for each arm respectively.
Measure: Number; unit: Participants
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 359 | 355
Participants
  Hemoglobin: Grade 1 (n =320, 316) | 93 | 112
  Hemoglobin: Grade 2 (n =320, 316) | 19 | 41
  Hemoglobin: Grade 3 (n =320, 316) | 1 | 11
  Hemoglobin: Grade 4 (n =320, 316) | 0 | 1
  Lymphocytes: Grade 1 (n =317, 309) | 7 | 7
  Lymphocytes: Grade 2 (n =317, 309) | 89 | 93
  Lymphocytes: Grade 3 (n =317, 309) | 10 | 11
  Lymphocytes: Grade 4 (n =317, 309) | 0 | 0
  Neutrophils: Grade 1 (n =316, 308) | 13 | 20
  Neutrophils: Grade 2 (n =316, 308) | 4 | 4
  Neutrophils: Grade 3 (n =316, 308) | 2 | 2
  Neutrophils: Grade 4 (n =316, 308) | 0 | 0
  Platelets: Grade 1 (n =312, 310) | 47 | 41
  Platelets: Grade 2 (n =312, 310) | 0 | 3
  Platelets: Grade 3 (n =312, 310) | 1 | 0
  Platelets: Grade 4 (n =312, 310) | 0 | 0
  White Blood Cells: Grade 1 (n =320, 315) | 32 | 36
  White Blood Cells: Grade 2 (n =320, 315) | 4 | 12
  White Blood Cells: Grade 3 (n =320, 315) | 0 | 1
  White Blood Cells: Grade 4 (n =320, 315) | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Biochemistry
Description: Biochemistry laboratory test included parameters: alanine aminotransferase, alkaline phosphatase, amylase, aspartate aminotransferase, bicarbonate, bilirubin, creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hyponatremia, hypophosphatemia and lipase. Abnormalities were assessed by CTCAE Grade Version 2 for severity: Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 359 | 355
Participants
  Alanine aminotransferase: Grade 1 (n =331, 313) | 65 | 57
  Alanine aminotransferase: Grade 2 (n =331, 313) | 8 | 6
  Alanine aminotransferase: Grade 3 (n =331, 313) | 1 | 2
  Alanine aminotransferase: Grade 4 (n =331, 313) | 0 | 3
  Alkaline phosphatase: Grade 1 (n =336, 319) | 88 | 92
  Alkaline phosphatase: Grade 2 (n =336, 319) | 8 | 15
  Alkaline phosphatase: Grade 3 (n =336, 319) | 4 | 3
  Alkaline phosphatase: Grade 4 (n =336, 319) | 0 | 0
  Amylase: Grade 1 (n =338, 319) | 64 | 76
  Amylase: Grade 2 (n =338, 319) | 12 | 21
  Amylase: Grade 3 (n =338, 319) | 7 | 6
  Amylase: Grade 4 (n =338, 319) | 0 | 1
  Aspartate aminotransferase: Grade 1 (n =331, 311) | 59 | 67
  Aspartate aminotransferase: Grade 2 (n =331, 311) | 5 | 7
  Aspartate aminotransferase: Grade 3 (n =331, 311) | 1 | 4
  Aspartate aminotransferase: Grade 4 (n =331, 311) | 0 | 0
  Bicarbonate: Grade 1 (n =314, 291) | 127 | 115
  Bicarbonate: Grade 2 (n =314, 291) | 11 | 10
  Bicarbonate: Grade 3 (n =314, 291) | 0 | 0
  Bicarbonate: Grade 4 (n =314, 291) | 1 | 0
  Bilirubin: Grade 1 (n =336, 318) | 16 | 12
  Bilirubin: Grade 2 (n =336, 318) | 8 | 2
  Bilirubin: Grade 3 (n =336, 318) | 1 | 1
  Bilirubin: Grade 4 (n =336, 318) | 0 | 0
  Creatinine: Grade 1 (n =336, 318) | 155 | 121
  Creatinine: Grade 2 (n =336, 318) | 30 | 9
  Creatinine: Grade 3 (n =336, 318) | 0 | 1
  Creatinine: Grade 4 (n =336, 318) | 0 | 0
  Hypercalcemia: Grade 1 (n =336, 319) | 92 | 22
  Hypercalcemia: Grade 2 (n =336, 319) | 8 | 1
  Hypercalcemia: Grade 3 (n =336, 319) | 1 | 0
  Hypercalcemia: Grade 4 (n =336, 319) | 0 | 0
  Hyperglycemia: Grade 1 (n =336, 319) | 41 | 28
  Hyperglycemia: Grade 2 (n =336, 319) | 45 | 37
  Hyperglycemia: Grade 3 (n =336, 319) | 7 | 7
  Hyperglycemia: Grade 4 (n =336, 319) | 0 | 0
  Hyperkalemia: Grade 1 (n =333, 314) | 0 | 0
  Hyperkalemia: Grade 2 (n =333, 314) | 42 | 22
  Hyperkalemia: Grade 3 (n =333, 314) | 9 | 8
  Hyperkalemia: Grade 4 (n =333, 314) | 0 | 0
  Hypernatremia: Grade 1 (n =338, 319) | 34 | 23
  Hypernatremia: Grade 2 (n =338, 319) | 19 | 14
  Hypernatremia: Grade 3 (n =338, 319) | 3 | 1
  Hypernatremia: Grade 4 (n =338, 319) | 0 | 2
  Hypoalbuminemia: Grade 1 (n =337, 319) | 37 | 25
  Hypoalbuminemia: Grade 2 (n =337, 319) | 11 | 31
  Hypoalbuminemia: Grade 3 (n =337, 319) | 1 | 2
  Hypoalbuminemia: Grade 4 (n =337, 319) | 0 | 0
  Hypocalcemia: Grade 1 (n =336, 319) | 25 | 67
  Hypocalcemia: Grade 2 (n =336, 319) | 4 | 18
  Hypocalcemia: Grade 3 (n =336, 319) | 2 | 2
  Hypocalcemia: Grade 4 (n =336, 319) | 1 | 2
  Hypoglycemia: Grade 1 (n =336, 319) | 23 | 9
  Hypoglycemia: Grade 2 (n =336, 319) | 12 | 16
  Hypoglycemia: Grade 3 (n =336, 319) | 1 | 1
  Hypoglycemia: Grade 4 (n =336, 319) | 0 | 0
  Hypokalemia: Grade 1 (n =333, 314) | 22 | 21
  Hypokalemia: Grade 2 (n =333, 314) | 0 | 0
  Hypokalemia: Grade 3 (n =333, 314) | 0 | 5
  Hypokalemia: Grade 4 (n =333, 314) | 0 | 0
  Hyponatremia: Grade 1 (n =338, 319) | 33 | 27
  Hyponatremia: Grade 2 (n =338, 319) | 0 | 0
  Hyponatremia: Grade 3 (n =338, 319) | 11 | 6
  Hyponatremia: Grade 4 (n =338, 319) | 1 | 1
  Hypophosphatemia: Grade 1 (n =336, 318) | 4 | 8
  Hypophosphatemia: Grade 2 (n =336, 318) | 33 | 99
  Hypophosphatemia: Grade 3 (n =336, 318) | 6 | 51
  Hypophosphatemia: Grade 4 (n =336, 318) | 0 | 0
  Lipase: Grade 1 (n =338, 319) | 53 | 76
  Lipase: Grade 2 (n =338, 319) | 22 | 25
  Lipase: Grade 3 (n =338, 319) | 14 | 40
  Lipase: Grade 4 (n =338, 319) | 2 | 7

10. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Urinalysis
Description: Urinalysis included urine blood/ hemoglobin, glucose and protein. Abnormalities were assessed by CTCAE Grade Version 2 for severity: Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 359 | 355
Participants
  Urine blood/ hemoglobin: Grade 1 (n =304, 272) | 45 | 35
  Urine blood/ hemoglobin: Grade 2 (n =304, 272) | 1 | 0
  Urine blood/ hemoglobin: Grade 3 (n =304, 272) | 0 | 0
  Urine blood/ hemoglobin: Grade 4 (n =304, 272) | 0 | 0
  Urine glucose: Grade 1 (n =322, 286) | 12 | 13
  Urine glucose: Grade 2 (n =322, 286) | 0 | 3
  Urine glucose: Grade 3 (n =322, 286) | 0 | 0
  Urine glucose: Grade 4 (n =322, 286) | 1 | 1
  Urine protein: Grade 1 (n =326, 289) | 105 | 91
  Urine protein: Grade 2 (n =326, 289) | 31 | 27
  Urine protein: Grade 3 (n =326, 289) | 27 | 21
  Urine protein: Grade 4 (n =326, 289) | 9 | 7

11. Secondary Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index-15 (FKSI-15) Score
Description: FKSI was used to assess quality of life (QoL) for those diagnosed with renal cell cancer and consisted of 15 items (lack of energy, side effects, pain, losing weight, bone pain, fatigue, enjoying life, short of breath, worsened condition, appetite, coughing, bothered by fevers, ability to work, hematuria and sleep). Each of the 15 items was answered on a 5-point Likert-type scale ranging from 0 to 4 (0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4= very much). Total FKSI score = sum of the 15 item scores; total range: 0 - 60; 0 (no symptoms) to 60 (very much); higher scores indicate greater presence of symptoms.
Time Frame: Baseline (Predose on Cycle 1 Day 1) , Day 1 of each cycle until Cycle 21, End of treatment (Day 670) and Follow-up visit (Day 698)
Population: FAS included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized. Here, "n" signifies those participants who were evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Units on a scale
  Baseline (n =346, 342) | 43.199 (8.416) | 43.339 (8.162)
  Cycle 2/Day1 (n =319, 296) | 42.351 (8.305) | 41.668 (7.696)
  Cycle 3/Day1 (n =279, 246) | 42.590 (7.729) | 42.424 (7.888)
  Cycle 4/Day1 (n =257, 221) | 42.791 (8.180) | 43.424 (7.345)
  Cycle 5/Day1 (n =238, 203) | 42.968 (8.152) | 42.907 (7.255)
  Cycle 6/Day1 (n =213, 179) | 42.949 (7.842) | 43.057 (7.724)
  Cycle 7/Day1 (n =206, 158) | 42.747 (7.621) | 43.578 (7.621)
  Cycle 8/Day1 (n =177, 136) | 43.580 (7.578) | 44.074 (7.757)
  Cycle 9/Day1 (n =163, 118) | 43.191 (8.300) | 44.518 (6.511)
  Cycle 10/Day1 (n =146, 96) | 43.312 (8.564) | 44.771 (7.155)
  Cycle 11/Day1 (n =122, 85) | 44.119 (8.306) | 44.438 (7.388)
  Cycle 12/Day1 (n =110, 70) | 44.517 (8.212) | 44.357 (7.247)
  Cycle 13/Day1 (n =92, 58) | 44.492 (7.972) | 45.261 (7.840)
  Cycle 14/Day1 (n =81, 54) | 44.485 (8.204) | 44.898 (7.495)
  Cycle 15/Day1 (n =61, 38) | 45.291 (7.095) | 45.053 (6.682)
  Cycle 16/Day1 (n =52, 34) | 45.217 (7.656) | 44.445 (7.160)
  Cycle 17/Day1 (n =47, 28) | 45.242 (7.344) | 44.438 (7.683)
  Cycle 18/Day1 (n =36, 22) | 44.861 (7.769) | 44.182 (7.228)
  Cycle 19/Day1 (n =29, 14) | 45.379 (6.662) | 45.026 (7.705)
  Cycle 20/Day1 (n =20, 12) | 47.050 (5.375) | 44.780 (6.689)
  Cycle 21/Day1 (n =15, 7) | 45.850 (5.209) | 44.494 (6.153)
  End of treatment (n=163, 191) | 38.328 (9.472) | 38.457 (8.787)
  Follow up (n =80, 110) | 41.919 (8.318) | 40.028 (9.048)

12. Secondary Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index-Disease Related Symptoms (FKSI-DRS) Score
Description: FKSI-DRS was used to assess quality of life for those diagnosed with renal cell cancer and consisted of 9 items (lack of energy, pain, losing weight, bone pain, fatigue, short of breath, coughing, bothered by fevers, and hematuria). Each of the 9 items was answered on a 5-point Likert-type scale ranging from 0 to 4 (0= not at all, 1= a little bit, 2= somewhat, 3= quite a bit, 4= very much). Total FKSI-DRS score = sum of the 9 item scores; total range: 0 - 36; 0 (no symptoms) to 36 (very much); higher scores indicate greater presence of symptoms.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Units on a scale
  Baseline (n =346, 341) | 28.874 (5.187) | 28.975 (5.193)
  Cycle 2/Day1 (n =319, 295) | 28.211 (4.920) | 28.399 (5.064)
  Cycle 3/Day1 (n =279, 244) | 28.640 (4.837) | 28.640 (4.868)
  Cycle 4/Day1 (n =257, 220) | 28.822 (4.952) | 29.130 (4.322)
  Cycle 5/Day1 (n =238, 202) | 28.869 (4.880) | 29.007 (4.379)
  Cycle 6/Day1 (n =213, 178) | 29.159 (4.462) | 29.098 (4.697)
  Cycle 7/Day1 (n =206, 157) | 29.042 (4.581) | 29.361 (4.558)
  Cycle 8/Day1 (n =177, 135) | 29.520 (4.346) | 29.619 (4.386)
  Cycle 9/Day1 (n =163, 117) | 29.194 (4.937) | 29.884 (3.838)
  Cycle 10/Day1 (n =146, 96) | 29.343 (4.907) | 29.604 (3.959)
  Cycle 11/Day1 (n =122, 85) | 29.762 (4.943) | 29.366 (4.404)
  Cycle 12/Day1 (n =110, 70) | 29.764 (4.507) | 29.257 (4.299)
  Cycle 13/Day1 (n =92, 58) | 29.594 (4.205) | 29.666 (4.710)
  Cycle 14/Day1 (n =81, 54) | 29.711 (4.313) | 29.820 (4.333)
  Cycle 15/Day1 (n =61, 38) | 30.324 (3.582) | 29.500 (3.454)
  Cycle 16/Day1 (n =52, 34) | 30.430 (3.443) | 29.474 (4.146)
  Cycle 17/Day1 (n =47, 28) | 30.551 (3.331) | 28.737 (4.930)
  Cycle 18/Day1 (n =36, 22) | 30.194 (3.992) | 29.045 (4.520)
  Cycle 19/Day1 (n =29, 14) | 30.130 (3.636) | 29.286 (4.795)
  Cycle 20/Day1 (n =20, 12) | 31.300 (2.736) | 29.250 (4.025)
  Cycle 21/Day1 (n =15, 7) | 31.067 (3.173) | 30.143 (4.100)
  End of Treatment (n =163, 191) | 26.288 (5.806) | 26.517 (5.614)
  Follow up (n =80, 110) | 28.263 (4.802) | 27.516 (5.577)

13. Secondary Outcome: Euro Quality of Life Questionnaire- 5 Dimension (EQ-5D): Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility or index score. Health state profile component assesses level of health for 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain was rated on a 3-point response scale (1= no problems, 2= some/moderate problems and 3= extreme problems). Scoring formula developed by EuroQol Group assigned a utility value for each domain in the profile. Score were transformed and resulted in a total score range of 0 to 1, with higher scores indicating better health.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Units on a scale
  Baseline (n =347, 341) | 0.732 (0.275) [lower limit 0.275] | 0.731 (0.257)
  Cycle 2/Day1 (n =326, 307) | 0.716 (0.267) | 0.696 (0.237)
  Cycle 3/Day1 (n =287, 248) | 0.722 (0.243) | 0.709 (0.239)
  Cycle 4/Day1 (n =262, 226) | 0.730 (0.236) | 0.716 (0.248)
  Cycle 5/Day1 (n =244, 207) | 0.730 (0.237) | 0.711 (0.243)
  Cycle 6/Day1 (n =221, 178) | 0.734 (0.230) | 0.704 (0.246)
  Cycle 7/Day1 (n =213, 163) | 0.718 (0.267) | 0.728 (0.228)
  Cycle 8/Day1 (n =181, 136) | 0.756 (0.236) | 0.702 (0.259)
  Cycle 9/Day1 (n =169, 120) | 0.760 (0.227) | 0.730 (0.229)
  Cycle 10/Day1 (n =151, 98) | 0.734 (0.243) | 0.730 (0.233)
  Cycle 11/Day1 (n =126, 87) | 0.764 (0.235) | 0.724 (0.250)
  Cycle 12/Day1 (n =110, 73) | 0.744 (0.244) | 0.734 (0.232)
  Cycle 13/Day1 (n =96, 61) | 0.760 (0.211) | 0.753 (0.232)
  Cycle 14/Day1 (n =80, 57) | 0.723 (0.239) | 0.752 (0.211)
  Cycle 15/Day1 (n =63, 41) | 0.730 (0.255) | 0.758 (0.191)
  Cycle 16/Day1 (n =54, 37) | 0.749 (0.220) | 0.785 (0.158)
  Cycle 17/Day1 (n =48, 29) | 0.779 (0.186) | 0.764 (0.193)
  Cycle 18/Day1 (n =37, 20) | 0.755 (0.204) | 0.755 (0.208)
  Cycle 19/Day1 (n =29, 14) | 0.734 (0.253) | 0.804 (0.184)
  Cycle 20/Day1 (n =21, 12) | 0.794 (0.220) | 0.771 (0.182)
  Cycle 21/Day1 (n =16, 7) | 0.700 (0.273) | 0.771 (0.182)
  End of Treatment (n =169, 196) | 0.608 (0.316) | 0.612 (0.310)
  Follow up (n =76, 106) | 0.682 (0.294) | 0.666 (0.295)

14. Secondary Outcome: Euro Quality of Life Questionnaire- 5 Dimension (EQ-5D): Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. VAS component: participants rated their current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Number analyzed (Participants) | 361 | 362
Units on a scale
  Baseline (n =341, 339) | 70.560 (19.187) [lower limit 0.275] | 70.351 (17.403)
  Cycle 2/Day1 (n =317, 302) | 69.003 (20.195) | 67.606 (18.265)
  Cycle 3/Day1 (n =280, 250) | 69.843 (17.927) | 69.712 (18.429)
  Cycle 4/Day1 (n =261, 224) | 69.180 (18.636) | 70.759 (17.189)
  Cycle 5/Day1 (n =244, 205) | 69.705 (18.330) | 71.888 (16.999)
  Cycle 6/Day1 (n =220, 178) | 69.900 (18.168) | 71.365 (17.019)
  Cycle 7/Day1 (n =209, 163) | 69.919 (18.063) | 72.282 (17.521)
  Cycle 8/Day1 (n =180, 139) | 70.756 (19.183) | 71.475 (18.523)
  Cycle 9/Day1 (n =168, 121) | 70.667 (18.556) | 73.380 (17.473)
  Cycle 10/Day1 (n =151, 98) | 70.629 (18.680) | 75.102 (14.854)
  Cycle 11/Day1 (n =126, 87) | 72.103 (18.064) | 74.586 (15.161)
  Cycle 12/Day1 (n =111, 73) | 71.730 (17.276) | 73.959 (15.852)
  Cycle 13/Day1 (n =94, 61) | 70.723 (19.147) | 75.693 (14.571)
  Cycle 14/Day1 (n =81, 58) | 69.420 (20.286) | 75.362 (15.875)
  Cycle 15/Day1 (n =62, 42) | 73.016 (15.325) | 75.357 (15.368)
  Cycle 16/Day1 (n =52, 37) | 70.269 (19.272) | 73.676 (15.699)
  Cycle 17/Day1 (n =48, 30) | 71.375 (17.840) | 73.767 (16.298)
  Cycle 18/Day1 (n =37, 23) | 70.459 (18.853) | 73.870 (16.904)
  Cycle 19/Day1 (n =29, 14) | 71.034 (16.963) | 70.571 (17.956)
  Cycle 20/Day1 (n =21, 12) | 73.143 (15.347) | 66.917 (17.758)
  Cycle 21/Day1 (n =16, 7) | 74.563 (16.054) | 64.714 (16.183)
  End of Treatment (n =166, 197) | 61.759 (21.668) | 61.690 (20.973)
  Follow up (n =76, 109) | 64.382 (21.392) | 66.037 (19.754)

ADVERSE EVENTS:
Time Frame: From initiation of treatment up to follow-up period (up to 3 years)
Description: Same event may appear as both AE and SAE, what is presented are distinct event. Event may be classified as serious in 1 participant, nonserious in other, or 1 participant may have experienced both serious, nonserious event during study.
Arm/Group | Axitinib 5 mg | Sorafenib 400 mg
Serious Adverse Events (participants affected / at risk) | 146/359 | 127/355
Other Adverse Events (participants affected / at risk) | 337/359 | 346/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Axitinib 5 mg (N=359) | Sorafenib 400 mg (N=355)
Anaemia (Blood and lymphatic system disorders) | 0 | 8
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Haemorrhage coronary artery (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 6 | 4
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Secondary hypothyroidism (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Retinal artery embolism (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 5
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 2 | 2
Chills (General disorders) | 1 | 0
Death (General disorders) | 3 | 6
Device dislocation (General disorders) | 0 | 1
Disease progression (General disorders) | 32 | 18
Fatigue (General disorders) | 4 | 0
General physical health deterioration (General disorders) | 3 | 5
Hernia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 2 | 3
Pyrexia (General disorders) | 7 | 5
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Budd-Chiari syndrome (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Aspergillus infection (Infections and infestations) | 0 | 1
Bacterial diarrhoea (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 4
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count abnormal (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 10 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0
Meningeal disorder (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/265 | 0/258 — This event was gender specific.
Menometrorrhagia (Reproductive system and breast disorders) | 0/96 | 1/104 — This event was gender specific.
Vaginal polyp (Reproductive system and breast disorders) | 1/96 | 0/104 — This event was gender specific.
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Pain management (Surgical and medical procedures) | 0 | 1
Vertebroplasty (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 4
Infarction (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib 5 mg (N=359) | Sorafenib 400 mg (N=355)
Anaemia (Blood and lymphatic system disorders) | 18 | 44
Hypothyroidism (Endocrine disorders) | 74 | 33
Abdominal pain (Gastrointestinal disorders) | 55 | 46
Abdominal pain upper (Gastrointestinal disorders) | 37 | 16
Constipation (Gastrointestinal disorders) | 79 | 82
Diarrhoea (Gastrointestinal disorders) | 208 | 195
Dyspepsia (Gastrointestinal disorders) | 39 | 15
Flatulence (Gastrointestinal disorders) | 20 | 8
Nausea (Gastrointestinal disorders) | 128 | 84
Stomatitis (Gastrointestinal disorders) | 60 | 47
Vomiting (Gastrointestinal disorders) | 95 | 69
Asthenia (General disorders) | 78 | 57
Chest pain (General disorders) | 23 | 20
Fatigue (General disorders) | 151 | 122
Mucosal inflammation (General disorders) | 61 | 45
Oedema peripheral (General disorders) | 22 | 22
Pain (General disorders) | 19 | 17
Pyrexia (General disorders) | 26 | 40
Nasopharyngitis (Infections and infestations) | 25 | 13
Blood thyroid stimulating hormone increased (Investigations) | 19 | 11
Lipase increased (Investigations) | 13 | 22
Weight decreased (Investigations) | 111 | 83
Decreased appetite (Metabolism and nutrition disorders) | 140 | 112
Dehydration (Metabolism and nutrition disorders) | 18 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 62 | 46
Back pain (Musculoskeletal and connective tissue disorders) | 59 | 54
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 21
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 28 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 | 53
Dizziness (Nervous system disorders) | 33 | 21
Dysgeusia (Nervous system disorders) | 43 | 31
Headache (Nervous system disorders) | 55 | 43
Insomnia (Psychiatric disorders) | 33 | 21
Proteinuria (Renal and urinary disorders) | 49 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 68 | 70
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 116 | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 64 | 53
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 | 19
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 21
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 122
Dry skin (Skin and subcutaneous tissue disorders) | 36 | 42
Erythema (Skin and subcutaneous tissue disorders) | 12 | 39
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 100 | 183
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 48
Rash (Skin and subcutaneous tissue disorders) | 53 | 109
Hypertension (Vascular disorders) | 156 | 107
Hypotension (Vascular disorders) | 19 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.